CLINICAL TRIAL: NCT04118413
Title: Bilateral Ultrasound Guided Low Thoracic Erector Spinae Plane Block for Postoperative Analgesia in Caesarean Delivery
Brief Title: Ultrasound Guided Bilateral Erector Spinae Plane Block in Caesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cigli Regional Training Hospital (Other)
Responsible Party: Principal Investigator, Hakan Aygün, Principal Investigator,, Cigli Regional Training Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESPB for CD
Record Dates: First submitted 2019-10-05; First posted 2019-10-08 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector spinae plane block (Experimental): Erector spinae plane block will be administrated to this group at end of the surgery under spinal anesthesia. An intravenous patient-controlled analgesia device within morphine will be given to the patients postoperatively and sheduled paracetamol will be given.
  Interventions: Other: erector spinae plane block
- Control Group (No Intervention): In this group, patients will receive only multimodal analgesic treatment including patient-controlled analgesia with morphine and sheduled paracetamol. No block will be performed.

INTERVENTIONS:
Other: erector spinae plane block — Erector espine plane block will be administrated bilaterally to this group at low thoracic level (Th11).
  Arms: Erector spinae plane block

SUMMARY:
Erector Spinae plane block (ESPB) is a regional anesthesia technique described three years ago. Its use for many indications has been identified by case reports in the literature. As the investigators have considered that ESPB could be efficacious for providing postoperative analgesia in the cesarean section, the investigators have implemented the application of this blockade into practice at the clinic. The main purpose of this study is to evaluate the analgesic effect of ultrasound-guided bilateral low thoracic ESPB in cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing cesarean section under spinal anesthesia

Exclusion Criteria:

* patients undergoing cesarean section under general anesthesia morbidly obesity, ASA III - IV , infection of the skin at the site of needle puncture area, patients with known allergies to any of the study drugs, coagulopathy, recent use of analgesic drugs

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2019-12-17 (Actual)

PRIMARY OUTCOMES:
24 hours opioid consumption | 24 hour
  morphine consumptions for both group will be recorded

SECONDARY OUTCOMES:
Numeric rating scale for postoperative pain intensity | 24 hour
  Changes in Numeric Rating Scale (NRS) at rest and on movement will be recorded at intervals. NRS is a unidimensional measure of pain intensity in adults. The NRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").

CONTACTS AND LOCATIONS:
Overall Officials: Aygun, Principal Investigator — izmir cigli regional hospital
Locations (1):
- Cigli regional research hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yamak Altinpulluk E, Garcia Simon D, Fajardo-Perez M. Erector spinae plane block for analgesia after lower segment caesarean section: Case report. Rev Esp Anestesiol Reanim (Engl Ed). 2018 May;65(5):284-286. doi: 10.1016/j.redar.2017.11.006. Epub 2018 Jan 17. English, Spanish. PMID 29352577
- [Result] Santonastaso DP, de Chiara A, Addis A, Mastronardi C, Pini R, Agnoletti V. Ultrasound guided erector spinae plane block for post-operative pain control after caesarean section. J Clin Anesth. 2019 Dec;58:45-46. doi: 10.1016/j.jclinane.2019.05.009. Epub 2019 May 7. No abstract available. PMID 31075624
- [Result] Aygun H, Thomas DT, Tulgar S. Comment to Santonastaso et al. 'J Clin Anesth 2019; 58: 45-46' and report of erector spinae plane block series in caesarean delivery patients. J Clin Anesth. 2020 Mar;60:4-5. doi: 10.1016/j.jclinane.2019.08.008. Epub 2019 Aug 16. No abstract available. PMID 31425897